CLINICAL TRIAL: NCT05481905
Title: The ENACT Trial: A Randomized, Double-blind, Placebo-controlled Adjunctive Treatment Trial to Evaluate the Efficacy and Safety of ENX-101 in Patients With Focal (Partial Onset) Seizures
Brief Title: ENACT: A Study of ENX-101 as Adjunctive Treatment in Patients With Focal Seizures
Acronym: ENACT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Engrail Therapeutics INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENX-101-005
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-07

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ENX-101 15mg daily (Experimental)
  Interventions: Drug: ENX-101
- ENX-101 30mg daily (Experimental)
  Interventions: Drug: ENX-101
- Placebo daily (Placebo Comparator)
  Interventions: Drug: ENX-101

INTERVENTIONS:
Drug: ENX-101 — Adjunctive treatment to current antiseizure medication

SUMMARY:
The ENACT trial is designed to evaluate the efficacy and safety of ENX-101 administered adjunctively to current therapy in reducing seizure frequency in patients diagnosed with focal (partial onset) epilepsy and treated with 1 to 4 antiseizure medications yet still experiencing seizures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 75 years, inclusive, at Screening
2. Diagnosed with focal (partial onset) epilepsy according to the International League Against Epilepsy (ILAE) 2017 classification of Epilepsy, as confirmed by the Epilepsy Study Consortium
3. Able to provide an imaging study(ies) [magnetic resonance imaging (MRI) scan strongly preferred yet computed tomography (CT) acceptable] obtained within the previous 10 years that can rule out a progressive cause of epilepsy
4. During the 3 months (84 days) immediately prior to Screening:

   * ≥ 3 observable focal onset seizures per 28-day period
   * <10 seizures per day
   * Any seizure-free interval no more than 21 days in length,
5. During the 8-week Baseline Period prior to Day 1:

   * ≥ 6 observable focal onset seizures
   * < 10 seizures per day
   * No seizure-free interval of ≥ 21 days,
6. Has been treated with antiseizure medications (ASMs) ≥ 2 years and currently being treated with:

   * One to 4 ASMs at stable doses for at least 28 days before Screening (not including the rescue medication)
   * Dose adjustments not expected during study

Exclusion Criteria:

1. EEG shows any pattern not consistent with focal etiology of seizures (e.g., generalized spike-wave)
2. Has history of focal onset seizures which involve subjective sensory or psychic phenomena without impairment of consciousness or awareness (formerly referred to as simple partial seizures without observable component) as their only seizure type
3. Has genetic/idiopathic generalized epilepsies or combined generalized and focal epilepsies, including a history of Lennox-Gastaut syndrome
4. Has history of seizures that occur at such a high frequency they cannot be reliably counted (e.g., repetitive, cluster seizures) within the year prior to Screening
5. Has history of psychogenic non-epileptic seizures
6. Has history of status epilepticus within two years prior to Screening
7. Treatment of epilepsy with ASM was initiated < 2 years prior to Screening
8. Ingested excluded concomitant medication within 5 half lives or 28 days (whichever is longer) prior to Screening
9. Had epilepsy surgery for tissue resection < 1 year prior to Screening or radiosurgery < 2 years prior to Screening
10. Had Vagus Nerve Stimulation (VNS), Deep Brain Stimulation (DBS), Responsive Neurostimulator System (RNS), or other neurostimulation for epilepsy device implanted or activated < 1 year prior to Screening, stimulation parameters have been stable for < 3 months, or battery life of unit not anticipated to extend for duration of trial
11. Initiated dietary therapy for epilepsy (e.g., ketogenic diet) < 3 months prior to Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of ENX-101 administered adjunctively with 1 to 4 antiseizure medications for the treatment of focal seizures | Day 1 to end of the Treatment Period (Day 56) compared to placebo
  The median percent change from baseline in 28-day focal seizure frequency (focal aware motor with observable component, focal impaired awareness, or focal to bilateral tonic-clonic seizures) compared to placebo

SECONDARY OUTCOMES:
To evaluate the efficacy of ENX-101 administered adjunctively with 1 to 4 antiseizure medications for the treatment of focal seizures | Treatment Period (Day 1 to Day 56) compared to placebo
  The responder rate defined as the percent of patients who experience a 50% or greater reduction from baseline in seizure frequency in the Treatment Period compared to placebo (designated as primary for the European Medicines Agency)
To evaluate the efficacy of ENX-101 | Treatment Period (Day 29 to Day 56) compared to placebo
  The percent of patients who are seizure free during the last 28 days of the Treatment Period
To evaluate the efficacy of ENX-101 | Treatment Period (Day 1 to Day 56) compared to placebo
  The percent of patients who are seizure free during the entire Treatment Period

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Rancho Research Institute at Rancho Los Amigos National Rehabilitation Center, Downey, California
  - University of Colorado, Aurora, Colorado
  - University of Florida Research Institute of Orlando, Gainesville, Florida
  - Royal Care Medical Research Corporation, Miami, Florida
  - University of Miami, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - S&G Research Center Corp., Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Comprehensive Neurology Clinic, Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - OSF HealthCare Illinois Neurological Institute, Peoria, Illinois
  - University of Kansas, Kansas City, Kansas
  - Saint Joseph Health System, Lexington, Kentucky
  - Maine Medical Partners Neurology, Scarborough, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Oakland University William Beaumont School of Medicine, Farmington Hills, Michigan
  - SRI International, Plymouth, Michigan
  - Advanced Clinical Research Center, Bridgeton, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Somnos Clinical Research/Neurology Associates, Lincoln, Nebraska
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Institute of Neurology and Neurosurgery at Saint Barnabas LLC, Livingston, New Jersey
  - Donald and Barbara Zucker School of Medicine at Hofstra/Northwell, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Atrium Health, Chapel Hill, North Carolina
  - Duke University School of Medicine, Durham, North Carolina
  - NeuroScience Research Center, LLC, Canton, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - DJL Clinical Research, Rock Hill, South Carolina
  - Mt. Olympus Medical Research, Sugar Land, Texas
  - University of Virginia, Charlottesville, Virginia